CLINICAL TRIAL: NCT01629589
Title: Immunogenicity of Adacel® and BOOSTRIX® Vaccines in Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Td551; U1111-1127-6774 (Other: WHO)
Record Dates: First submitted 2012-06-22; First posted 2012-06-27 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Tetanus; Diphtheria; Pertussis; Whooping Cough
Keywords: Adacel® vaccine; Tetanus; Diphtheria; whooping cough; Pertussis; BOOSTRIX® vaccine
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — Tetanus Toxoid; adacel; Boostrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adacel® Vaccine Group (Experimental): Participants randomized to receive a single dose of Adacel® vaccine
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Adacel®)
- Boostrix® Vaccine Group (Active Comparator): Participants randomized to receive a single dose of Boostrix® vaccine
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine, Adsorbed (BOOSTRIX®)

INTERVENTIONS:
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Adacel®) — 0.5 mL, Intramuscular
  Other Names: Adacel®
  Arms: Adacel® Vaccine Group
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine, Adsorbed (BOOSTRIX®) — 0.5 mL, Intramuscular
  Other Names: BOOSTRIX®
  Arms: Boostrix® Vaccine Group

SUMMARY:
The aim of this study is to describe immunogenicity of a single booster dose of Adacel vaccine versus Boostrix vaccine among approximately 420 adolescents 11 to <13 years of age.

Primary objective:

* To describe seroprotection rates against tetanus and diphtheria in subjects randomized to receive either Adacel or Boostrix vaccine.

Observational objectives:

* To describe pre- and post-vaccination tetanus, diphtheria, and pertussis geometric mean antibody concentrations (GMCs) in subjects randomized to receive either Adacel or Boostrix vaccine.
* To describe booster response rates against tetanus, diphtheria, and pertussis in subjects randomized to receive either Adacel or Boostrix vaccine.
* To describe the rates of adverse events (AEs) immediately post-vaccination, and the rates of unsolicited AEs and serious adverse events (SAEs) following vaccination with Adacel or Boostrix vaccine from Visit 1 through Visit 2.

DETAILED DESCRIPTION:
Participants will be randomized in a 1:1 ratio to receive either Adacel or Boostrix vaccine.

Subjects will be monitored for immediate reactions for 15 minutes post-vaccination. Unsolicited adverse events and serious adverse events will be collected from Visit 1 through Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 11 to < 13 years of age at the time of vaccination
* Received exactly 5 doses of pertussis vaccine at < 7 years of age
* Informed consent and assent forms have been signed and dated
* Subject is able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of child bearing potential without using an effective method of contraception or not practicing abstinence for at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination
* Any condition that, in the opinion of the Investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) within the past 3 months)
* Known or suspected receipt of any whole-cell pertussis-containing vaccine
* A personal history of physician-diagnosed or laboratory-confirmed pertussis disease within the last 2 years
* A previous severe reaction to pertussis, diphtheria or tetanus vaccine including immediate anaphylaxis, encephalopathy within 7 days, or seizure within 3 days of receiving the vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Suspected or known hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before the 2nd visit; except that influenza vaccine may have been received between 30 and 15 days (but no less than 15 days) before receiving study vaccine
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study, at the discretion of the Sponsor
* Seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C, as reported by the subject's parent/guardian
* Laboratory-confirmed thrombocytopenia, which may be a contraindication for intramuscular (IM) vaccination, at the discretion of the Investigator
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for IM vaccination, at the discretion of the Investigator
* Personal history of Guillain-Barré syndrome
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of vaccination. (A prospective subject should not be enrolled in the study until the condition has resolved or the febrile event has subsided.)
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol or drug use that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 423 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (8):
- United States (8):
  - Sacramento, California
  - Bardstown, Kentucky
  - Woburn, Massachusetts
  - Cleveland, Ohio
  - Barnwell, South Carolina
  - Kingsport, Tennessee
  - Salt Lake City, Utah
  - Vienna, Virginia

REFERENCES:
- [Derived] Decker MD, Greenberg DP, Johnson DR, Pool V. Randomized study of immune responses to two Tdap vaccines among adolescents primed with DTaP and comparison with results among adolescents primed with DTwP. Vaccine. 2019 Aug 14;37(35):5003-5008. doi: 10.1016/j.vaccine.2019.07.015. Epub 2019 Jul 10. PMID 31301919
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 20 June 2012 to 10 September 2012 at 8 centers in the United States.
Pre-assignment Details: A total of 423 participants that met all of the inclusion and none of the exclusion criteria were randomized, 422 were vaccinated in this study.
Groups:
- Adacel® Vaccine Group: Participants received a single dose of Adacel® vaccine
- BOOSTRIX® Vaccine Group: Participants received a single dose of BOOSTRIX® vaccine
Period: Overall Study
Arm/Group | Adacel® Vaccine Group | BOOSTRIX® Vaccine Group
Started | 212 | 211
Completed | 204 (A participant received the Boostrix vaccine. Study data reported for the Boostrix vaccine group.) | 204
Not Completed | 8 | 7
Not completed — Protocol Violation | 4 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Did not receive study vaccine | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adacel® Vaccine Group | BOOSTRIX® Vaccine Group | Total
Number analyzed (Participants) | 212 | 211 | 423
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 212 | 211 | 423
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.6 (0.5) | 11.6 (0.5) | 11.6 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 106 | 211
  Male | 107 | 105 | 212
Region of Enrollment [Number; unit: Participants]
  United States | 212 | 211 | 423

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Antibody Responses to Tetanus and Diphtheria Components Following Vaccination With Either Adacel® or BOOSTRIX® Vaccine
Description: Tetanus antibody was assayed by Enzyme-linked immunosorbent assay (ELISA) and Diphtheria antibody by a toxin neutralization test. Antibody responses to tetanus and diphtheria components were defined as titers ≥0.1 IU/mL and ≥1.0 IU/mL
Time Frame: Day 0 (pre-vaccination) to Day 28 (post-vaccination)
Population: The antibody responses to tetanus and diphtheria components were determined in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Adacel® Vaccine Group | BOOSTRIX® Vaccine Group
Number analyzed (Participants) | 196 | 194
Participants
  Tetanus (pre-vaccination) ≥0.1 IU/mL | 172 | 177 [0 to 0]
  Tetanus (post-vaccination) ≥0.1 IU/mL | 196 | 194 [0 to 0]
  Diphtheria (pre-vaccination) ≥0.1 IU/mL | 135 | 139 [0 to 0]
  Diphtheria (post-vaccination) ≥ 0.1 IU/mL | 196 | 194 [0 to 0]
  Tetanus (pre-vaccination) ≥ 1.0 IU/mL | 33 | 48 [0 to 0]
  Tetanus (post-vaccination) ≥ 1.0 IU/mL | 195 | 194 [0 to 0]
  Diphtheria (pre-vaccination) ≥1.0 IU/mL | 28 | 26 [0 to 0]
  Diphtheria (post-vaccination) ≥1.0 IU/mL | 183 | 186 [0 to 0]

2. Secondary Outcome: Geometric Mean Concentrations of Tetanus and Diphtheria Antibodies Following Vaccination With Either Adacel® or BOOSTRIX® Vaccine
Description: Tetanus antibody was assayed by Enzyme-linked immunosorbent assay (ELISA) and Diphtheria antibody by a toxin neutralization test
Time Frame: Day 0 (pre-vaccination) to Day 28 post-vaccination
Population: The geometric mean concentrations of tetanus and diphtheria antibodies were determined in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Adacel® Vaccine Group | BOOSTRIX® Vaccine Group
Number analyzed (Participants) | 196 | 194
Titers
  Tetanus (pre-vaccination) | 0.422 [0.363 to 0.492] | 0.456 [0.393 to 0.528]
  Tetanus (post-vaccination) | 18.9 [16.4 to 21.8] | 9.18 [8.10 to 10.4]
  Diphtheria (pre-vaccination) | 0.211 [0.171 to 0.260] | 0.221 [0.181 to 0.269]
  Diphtheria (post-vaccination) | 8.17 [6.83 to 9.77] | 5.62 [4.85 to 6.51]

3. Secondary Outcome: Number of Participants With Booster Responses Against Tetanus and Diphtheria Antigens Following Vaccination With Either Adacel® or BOOSTRIX® Vaccine
Description: Adacel booster response defined as: a 4-fold increase in pre- to post-vaccination antibody concentrations for subjects with a pre-vaccination concentration ≤2.56 IU/mL for diphtheria and ≤2.7 IU/mL for tetanus, and defined as a 2-fold increase for subjects with a pre-vaccination concentration >2.56 IU/mL for diphtheria and >2.7 IU/mL for tetanus.
  Boostrix booster response defined as: a post-vaccination titer ≥4 times the lower limit of quantitation (LLOQ) for subjects with a pre-vaccination titer < LLOQ, a post-vaccination titer ≥4 times the pre-vaccination titer for subjects with a pre-vaccination titer between LLOQ and 4x LLOQ, or a post-vaccination titer at least twice the pre-vaccination titer for subjects with a pre-vaccination titer ≥4x LLOQ.
Time Frame: Day 28 post-vaccination
Population: Booster response against tetanus and diphtheria components were determined in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Adacel® Vaccine Group | BOOSTRIX® Vaccine Group
Number analyzed (Participants) | 196 | 194
Participants
  Tetanus | 194 | 191
  Diphtheria | 189 | 188

4. Secondary Outcome: Geometric Mean Concentrations of the Pertussis Antibodies Following Vaccination With Either Adacel® or BOOSTRIX® Vaccine
Description: Pertussis antibodies Pertussis toxoid (PT), Filamentous hemagglutinin (FHA), Pertactin (PRN), and Fimbriae types 2 and 3 (FIM 2&3) were assayed by Enzyme-linked immunosorbent assay (ELISA)
Time Frame: Day 0 (pre-vaccination) to Day 28 post-vaccination
Population: Geometric mean concentrations of the Pertussis antibodies were determined in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Adacel® Vaccine Group | BOOSTRIX® Vaccine Group
Number analyzed (Participants) | 196 | 194
Titers
  Pertussis toxoid (pre-vaccination) | 5.59 [4.67 to 6.68] | 5.69 [4.71 to 6.88]
  Pertussis toxoid (post-vaccination) | 31.0 [27.0 to 35.7] | 44.1 [39.0 to 49.9]
  Filamentous hemagglutinin (pre-vaccination) | 22.7 [19.0 to 27.2] | 22.7 [19.4 to 26.6]
  Filamentous hemagglutinin (post-vaccination) | 255 [228 to 286] | 318 [292 to 347]
  Pertactin (pre-vaccination) | 12.3 [10.5 to 14.4] | 10.3 [8.99 to 11.9]
  Pertactin (post-vaccination) | 263 [223 to 310] | 252 [214 to 295]
  Fimbriae types 2 and 3 (pre-vaccination) | 5.95 [4.88 to 7.24] | 6.55 [5.33 to 8.04]
  Fimbriae types 2 and 3 (post-vaccination) | 346 [269 to 446] | 11.1 [8.79 to 14.0]

5. Secondary Outcome: Number of Participants With Booster Responses Against the Pertussis Antibodies Following Vaccination With Either Adacel® or BOOSTRIX® Vaccine
Description: Adacel booster response defined as: a 4-fold increase in pre- to post-vaccination antibody concentrations for subjects with a pre vaccination concentration ≤93 ELISA Unit (EU)/mL for Pertussis toxoid (PT), ≤170 EU/mL for Filamentous hemagglutinin (FHA), ≤115 EU mL for pertactin (PRN), or ≤285 EU/mL for Fimbriae types 2 and 3 (FIM), and defined as a 2-fold increase for subjects with a pre-vaccination concentration >93 EU/mL for PT, >170 EU/mL for FHA, >115 EU/mL for PRN, or >285 EU/mL for FIM.
  Boostrix booster response defined as: a post-vaccination titer ≥4 times the LLOQ for subjects with a pre-vaccination titer <LLOQ, a post-vaccination titer ≥4 times the pre-vaccination titer for subjects with a pre-vaccination titer between LLOQ and 4x LLOQ, or a post-vaccination titer at least twice the pre-vaccination titer for subjects with a pre-vaccination titer ≥4x LLOQ.
Time Frame: Day 28 post-vaccination
Population: Booster response against Pertussis antibodies were determined in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Adacel® Vaccine Group | BOOSTRIX® Vaccine Group
Number analyzed (Participants) | 196 | 194
Participants
  Pertussis toxoid | 97 [45.2 to 60.1] | 142 [0 to 0]
  Filamentous hemagglutinin | 167 [79.4 to 89.9] | 189 [0 to 0]
  Pertactin | 186 [90.8 to 97.5] | 189 [0 to 0]
  Fimbriae types 2 and 3 | 181 [87.7 to 95.7] | 31 [0 to 0]

6. Secondary Outcome: Number of Participants Reporting Immediate Unsolicited Adverse Events Following Vaccination With Either Adacel® or BOOSTRIX® Vaccine
Description: The occurrence, nature (Medical Dictionary for Regulatory Activities (MedDRA) preferred term), duration, intensity, and relationship to vaccination of adverse events (AEs) reported in the 15 minutes after vaccination and systemic AEs.
Time Frame: Up to 15 minutes post-vaccination
Population: Number of participants reporting immediate unsolicited adverse events was determined in all participants in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Adacel® Vaccine Group | BOOSTRIX® Vaccine Group
Number analyzed (Participants) | 211 | 211
Participants
  Headache | 1 | 0 [0 to 0]
  Nausea | 1 | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to Day 28 post-vaccination.
Arm/Group | Adacel® Vaccine Group | BOOSTRIX® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/211 | 0/211
Other Adverse Events (participants affected / at risk) | 58/211 | 70/211
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adacel® Vaccine Group (N=211) | BOOSTRIX® Vaccine Group (N=211)
Injection Site Pain (General disorders) | 34 (36) | 43 (46)
Headache (Nervous system disorders) | 21 (26) | 31 (39)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications